CLINICAL TRIAL: NCT01091454
Title: Phase II Trial of Brostallicin and Cisplatin in Patients With Metastatic Triple Negative Breast Cancer
Brief Title: Brostallicin and Cisplatin in Treating Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N0937; NCCTG-N0937; CDR0000665441 (Registry Identifier: PDQ (Physician Data Query)); NCI-2011-02016 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2010-03-18; First posted 2010-03-24 (Estimated); Results first posted 2017-03-20 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-04

CONDITIONS: Triple-negative Breast Cancer
Keywords: stage IV breast cancer; triple-negative breast cancer; male breast cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms; Breast Neoplasms, Male | interventions — brostallicin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (cisplatin and brostallicin) (Experimental): Patients receive cisplatin IV over 2 hours on day 1 and brostallicin IV over 10 minutes on day 2. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: brostallicin; Drug: cisplatin

INTERVENTIONS:
Drug: brostallicin — Given IV
Drug: cisplatin — Given IV

SUMMARY:
This phase II trial studies how well brostallicin and cisplatin work in treating patients with breast cancer that has spread to other parts of the body (metastatic) and does not have estrogen receptors, progesterone receptors, or large amounts of human epidermal growth factor receptor 2 (HER2) on its cells (triple-negative). Drugs used in chemotherapy, such as brostallicin and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify any clinical efficacy of brostallicin and cisplatin in the treatment of breast cancer patients having a triple negative (estrogen receptor [ER]/progesterone receptor [PR]/HER2 negative) phenotype, as measured by progression-free survival (PFS) at 3 months.

SECONDARY OBJECTIVES:

I. To describe the confirmed tumor response rate of patients with measurable disease receiving brostallicin and cisplatin.

II. To describe the duration of response in patients with measurable disease receiving brostallicin and cisplatin.

III. To describe the 6-month progression-free survival of patients receiving brostallicin and cisplatin.

IV. To describe the overall survival (OS) of patients receiving brostallicin and cisplatin.

V. To evaluate the adverse event profile of the study regimen (adverse events graded using the Cancer Therapy Evaluation Program [CTEP] Active Version of the Common Terminology Criteria for Adverse Events [CTCAE]).

OUTLINE:

Patients receive cisplatin intravenously (IV) over 2 hours on day 1 and brostallicin IV over 10 minutes on day 2. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months until disease progression and then every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria

* Histologically or cytologically confirmed adenocarcinoma of the breast with clinical evidence of metastatic disease
* Triple negative breast cancer defined as HER2-(according to current American Society of Clinical Oncology [ASCO] College of American Pathologists [CAP] guidelines), ER- (defined as =< 1% by IHC) and PgR- (defined as =< 1% by IHC)
* 0 to 4 prior chemotherapy regimens in the metastatic setting
* Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Hemoglobin >= 10.0 g/dL
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Platelet count >= 100,000/mL
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Serum creatinine =< 1.5 mg/dL
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) and serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 3 x ULN or SGOT (AST) and SGPT (ALT) =< 5 x ULN if elevations are due to liver metastases
* Alkaline phosphatase =< 2.5 x ULN or alkaline phosphatase =< 5 x ULN if elevations are due to liver metastases
* Electrocardiogram (EKG) completed =< 15 days prior to registration
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1 or 2
* Life expectancy > 3 months
* Has written informed consent
* Willingness to return to NCCTG enrolling institution for treatment and follow-up
* Patient willing to provide blood samples for research purposes

Exclusion Criteria

* HER2 positive (3+ by IHC or fluorescence in situ hybridization [FISH] amplified) breast cancer by ASCO/CAP guidelines
* Estrogen receptor (ER) and/or progesterone receptor (PR/PgR) positive breast cancer (defined as > 1% of either receptor by IHC)
* Any of the following

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception (as determined by the treating physician) while on this study and for 30 days after end of treatment with the study drugs
* Stage III or IV invasive non-breast malignancy in =< 5 years prior to registration
* Pre-existing peripheral neuropathy of grade >= 2 (using the CTEP active version of the CTCAE)
* Major surgery =< 4 weeks prior to registration
* Chemotherapy or immunologic therapy =< 3 weeks prior to registration
* Radiotherapy =< 2 weeks prior to registration, except if to a non-target lesion only

  * NOTES:
  * Prior radiation to a target lesion is permitted only if there has been clear progression of the lesion since radiation was completed
  * If patient receives single dose radiation for palliation or radiation to non-target lesion, they may immediately proceed to registration without waiting 2 weeks
  * Acute adverse events from radiation must have resolved to =< grade 1 (according to the CTEP active version of the CTCAE)
* Evidence of active brain metastasis including leptomeningeal involvement

  * NOTE: Central nervous system (CNS) metastasis controlled by prior surgery and/or radiotherapy is allowed; to be considered controlled, there must be at least 2 months of no symptoms or evidence of progression prior to study entry and corticosteroid therapy given to control brain edema must have been discontinued
* History of allergy or hypersensitivity to the drugs used in this study (or their excipients) including platinum compounds (cisplatin, carboplatin)
* Active, unresolved infection
* Uncontrolled intercurrent illness including, but not limited to psychiatric illness/social situations or co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or would interfere significantly with the proper assessment of safety of the prescribed regimens or would limit compliance with study requirements or would make it undesirable for patient to participate in the trial
* Clinically significant cardiovascular or cerebrovascular disease, including any history of the following =< 6 months prior to registration:

  * Myocardial infarction
  * Unstable angina
  * New York Heart Association (NYHA) class II or greater congestive heart failure
  * Uncontrolled or clinically significant cardiac arrhythmia (patients with controlled atrial fibrillation are eligible)
* Currently receiving treatment in a different clinical study in which investigational procedures are performed or investigational therapies are administered

  * NOTE: Patient may not enroll in such clinical trials while participating in this study; exception may be granted for trials related to symptom management (cancer control) which do not employ hormonal treatments or treatments that may block the path of the targeted agents used in this trial
* Immunocompromised patients (other than that related to the use of corticosteroids) including patients known to be human immunodeficiency virus (HIV) positive with an acquired immune deficiency syndrome (AIDS)-defining illness; HIV positive patients with cluster of differentiation (CD)4 count within institutional normal range and no history of an AIDS-defining illness are eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2012-06 (Actual); Study Completion 2014-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alvaro Moreno Aspitia, MD, Study Chair — Mayo Clinic
Locations (266):
- United States (266):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Lusitana, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - Hawaii Medical Center - East, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Kauai Medical Clinic, Lihue, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Illinois CancerCare - Galesburg, Galesburg, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Moline, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - OSF Holy Family Medical Center, Monmouth, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Bettendorf, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - Mercy Cancer Center - West Lakes, Clive, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Alexandria, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Goldschmidt Cancer Center, Jefferson City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Comprehensive Cancer Care, PC, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Presbyterian Cancer Treatment Center at Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Wood County Oncology Center, Bowling Green, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Community Cancer Center, Elyria, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Southern Ohio Medical Center Cancer Center, Portsmouth, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - United States Air Force Medical Center - Wright-Patterson, Wright-Patterson Air Force Base, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Marshfield Clinic - Chippewa Center, Chippewa Falls, Wisconsin
  - Center for Cancer Treatment & Prevention at Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - St. Nicholas Hospital, Sheboygan, Wisconsin
  - Marshfield Clinic at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Cisplatin and Brostallicin): Patients receive 50 mg/m^2 cisplatin IV over 2 hours on day 1 and 10 mg/m^2 brostallicin IV over 10 minutes on day 2. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment (Cisplatin and Brostallicin)
Started | 48
Completed | 47
Not Completed | 1
Not completed — Ineligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Cisplatin and Brostallicin)
Number analyzed (Participants) | 47
Age, Continuous [Median (Full Range); unit: years] | 57 [34 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 47

OUTCOME MEASURES:

1. Primary Outcome: 3-month Progression-free Survival (3-mo PFS) Rate
Description: A patient is considered to be a 3-month progression-free survivor if the patient is on study treatment 3 months from registration without a documentation of disease progression. The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients and 95% confidence intervals for the true success proportion will be calculated according to the approach of Duffy and Santner. If some patients are lost to follow-up not having been observed for at least 3 months, an estimate and confidence interval for the 3-month PFS rate incorporating censoring will be computed using the method of Kaplan-Meier. Progression is defined using the revised RECIST guideline (v1.1) as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: 3 months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Treatment (Cisplatin and Brostallicin)
Number analyzed (Participants) | 47
proportion of participants | 0.511 [0.386 to 0.676]

2. Secondary Outcome: Confirmed Response Rate
Description: A confirmed response is defined to be either a CR or PR noted as the objective status on 2 consecutive evaluations at least 6 weeks apart. All patients meeting the eligibility criteria who have signed a consent form and have begun treatment will be evaluable for response. The confirmed response rate will be estimated by the number of confirmed responses in evaluable patients with measurable disease divided by the total number of evaluable patients with measurable disease. The appropriate confidence interval will be calculated. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <1 cm.; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 5 years
Population: Out of the total number of participants who completed the study and were evaluable for the primary endpoint and adverse events (as provided in the Participant Flow), only a subset of participants (Overall Number of Participants Analyzed specified above) were evaluable for the Confirmed Response Rate.
Measure: Number (95% Confidence Interval); unit: percentage of confirmed responses
Arm/Group | Treatment (Cisplatin and Brostallicin)
Number analyzed (Participants) | 45
percentage of confirmed responses | 22 [11 to 37]

3. Secondary Outcome: Duration of Response
Description: Duration of response is defined for all evaluable patients with measurable disease who have achieved a confirmed response as the date at which the patient's earliest best objective status is first noted to be either a CR or PR to the earliest date progression is documented. If a patient dies subsequent to the confirmed response without a documentation of disease progression, the patient will be considered to have had disease progression at the time of their death. The distribution of duration of response will be estimated using the method of Kaplan-Meier. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <1 cm.; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Cisplatin and Brostallicin)
Number analyzed (Participants) | 47
months | 4 [2.6 to 14.5]

4. Secondary Outcome: 6-month Progression-free Survival (6-mo PFS) Rate
Description: 6-month progression-free survival. A patient is considered to be a 6-month progression-free survivor if the patient is on study treatment 6 months from registration without a documentation of disease progression. The 6-month progression-free survival rate incorporating censoring will be computed using the method of Kaplan-Meier. Progression is defined using the revised RECIST guideline (v1.1) as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: At 6 months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Treatment (Cisplatin and Brostallicin)
Number analyzed (Participants) | 47
proportion of participants | 0.277 [0.174 to 0.439]

5. Secondary Outcome: Time to Disease Progression
Description: Time to disease progression is defined as the time from registration to the earliest date of documentation of disease progression. If a patient dies without a documentation of disease progression the patient will be considered to have had disease progression at the time of their death. If the patient is declared to be a major treatment violation, the patient will be censored on the date the treatment violation was declared to have occurred. The distribution of time to progression will be estimated using the method of Kaplan-Meier. Progression is defined using the revised RECIST guideline (v1.1) as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Cisplatin and Brostallicin)
Number analyzed (Participants) | 47
months | 3.2 [2.2 to 4.2]

6. Secondary Outcome: Survival Time
Description: Survival time is defined as the time from registration to death due to any cause. The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time Frame: Up to 5 years
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Treatment (Cisplatin and Brostallicin)
Number analyzed (Participants) | 47
months | 8.3 [4.7 to 14.9]

ADVERSE EVENTS:
Time Frame: Adverse events are assessed 15 days prior to registration and during the Active Monitoring Phase: once per cycle (<=3 days prior to each subsequent cycle) of treatment and at the end of treatment; for up to 5 years.
Description: This study will utilize the CTEP Active Version of NCI Common Terminology Criteria for Adverse Events (CTCAE) for adverse event monitoring and reporting (Version 4). All eligible patients that have initiated treatment will be considered evaluable for adverse event analyses. Adverse events will be graded using the NCI CTCAE coding scheme. The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine adverse event patterns.
Arm/Group | Treatment (Cisplatin and Brostallicin)
Serious Adverse Events (participants affected / at risk) | 29/48
Other Adverse Events (participants affected / at risk) | 48/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Cisplatin and Brostallicin) (N=48)
Anemia (Blood and lymphatic system disorders) | 4 (4)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 (7)
Atrial fibrillation (Cardiac disorders) | 1 (2)
Pericardial effusion (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Death NOS (General disorders) | 1 (1)
Fatigue (General disorders) | 3 (5)
Allergic reaction (Immune system disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 19 (19)
Platelet count decreased (Investigations) | 20 (24)
White blood cell decreased (Investigations) | 5 (5)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Cisplatin and Brostallicin) (N=48)
Anemia (Blood and lymphatic system disorders) | 35 (146)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (4)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2)
Pericardial effusion (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 4 (6)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 4 (5)
Eye disorders - Other, specify (Eye disorders) | 1 (1)
Watering eyes (Eye disorders) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Anal pain (Gastrointestinal disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 12 (23)
Diarrhea (Gastrointestinal disorders) | 17 (32)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (2)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 8 (8)
Nausea (Gastrointestinal disorders) | 30 (80)
Oral pain (Gastrointestinal disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 11 (22)
Chills (General disorders) | 1 (1)
Edema limbs (General disorders) | 3 (7)
Fatigue (General disorders) | 45 (189)
Fever (General disorders) | 3 (3)
Gait disturbance (General disorders) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1)
Infusion related reaction (General disorders) | 1 (1)
Localized edema (General disorders) | 2 (2)
Malaise (General disorders) | 2 (2)
Non-cardiac chest pain (General disorders) | 3 (4)
Pain (General disorders) | 3 (6)
Allergic reaction (Immune system disorders) | 6 (8)
Lung infection (Infections and infestations) | 1 (1)
Lymph gland infection (Infections and infestations) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 2 (5)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 7 (10)
Alkaline phosphatase increased (Investigations) | 23 (66)
Aspartate aminotransferase increased (Investigations) | 9 (15)
Blood bilirubin increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 10 (26)
GGT increased (Investigations) | 1 (1)
Hemoglobin increased (Investigations) | 2 (5)
Lymphocyte count decreased (Investigations) | 8 (24)
Neutrophil count decreased (Investigations) | 23 (43)
Platelet count decreased (Investigations) | 36 (105)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 2 (5)
White blood cell decreased (Investigations) | 16 (27)
Anorexia (Metabolism and nutrition disorders) | 6 (16)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (11)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (8)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (8)
Hypocalcemia (Metabolism and nutrition disorders) | 8 (14)
Hypokalemia (Metabolism and nutrition disorders) | 9 (15)
Hypomagnesemia (Metabolism and nutrition disorders) | 9 (20)
Hyponatremia (Metabolism and nutrition disorders) | 6 (15)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 5 (10)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (6)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (5)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 6 (8)
Dysgeusia (Nervous system disorders) | 5 (12)
Headache (Nervous system disorders) | 7 (12)
Memory impairment (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 7 (13)
Peripheral sensory neuropathy (Nervous system disorders) | 24 (95)
Syncope (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3)
Depression (Psychiatric disorders) | 1 (3)
Insomnia (Psychiatric disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (4)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 3 (5)
Vaginal dryness (Reproductive system and breast disorders) | 1 (3)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14 (33)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (8)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 12 (31)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (4)
Flushing (Vascular disorders) | 2 (2)
Hot flashes (Vascular disorders) | 1 (6)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (3)
Lymphedema (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes